CLINICAL TRIAL: NCT02821728
Title: A Pre-Biopsy Window of Opportunity Trial to Measure Sulphate Levels in Human Prostate After Broccoli Consumption
Brief Title: Sulphate Accumulation in Prostate
Acronym: SAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IFR01/2016
Record Dates: First submitted 2016-06-21; First posted 2016-07-04 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: Prostate; Sulphate; ATP; PTEN
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal diet (Experimental): No dietary intervention
  Interventions: Other: Normal diet
- Dietary intervention (Experimental): 3 portions of broccoli soup per week
  Interventions: Dietary Supplement: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary intervention — Participants in this group will consume three portions of broccoli and stilton soup per week for a minimum of four weeks before their scheduled template prostate biopsy. The soup will be made with a specially cultivated broccoli known as Beneforte, which contains an enhanced dose of a substance called glucoraphanin.
  Arms: Dietary intervention
Other: Normal diet — Participants in this group will continue with their normal diet up until the day of their scheduled template prostate biopsy.
  Arms: Normal diet

SUMMARY:
This study evaluates whether a broccoli intervention (≥ 4 weeks) will result in differences in tissue sulphate levels in men scheduled for prostate biopsies. Comparisons will be made between participants randomised to the broccoli-rich diet and those randomised to the non-intervention arm.

DETAILED DESCRIPTION:
Epidemiological studies provide evidence for a negative correlation between prostate cancer and intake of cruciferous vegetables such as broccoli. Preliminary data from ongoing intervention trials carried out at the IFR suggest that dietary changes can directly influence the metabolic profile of prostate tissue. The most significant result observed to date is that of sulphate accumulation within the prostate. The additional sulphate is likely to drive synthesis of 3'-phosphoadenosine-5'-phosphosulfate, a universal sulphate donor, a process which would consume energy from ATP. A significant rise in levels of both ADP and phosphate has also been observed in prostate tissue from these studies, supporting the potential depletion of cellular ATP. Interestingly, the data indicate that the extent of ADP accumulation is negatively correlated with prostate cancer progression.

The investigators now propose to undertake a two arm parallel un-blinded study to test the hypothesis that a short-term intervention with broccoli soups will lead to the accumulation of sulphate and ADP in prostate tissue. A potential increase in glutathione metabolites indicating a change in redox status, and therefore functional status, of specific genes involved in tumour suppression (PTEN) will also be investigated.

Furthermore, the investigators aim to determine whether the accumulation of sulphate and ADP is specific to the prostate gland through the metabolic analyses of both prostate and non-prostate tissues.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Scheduled for TPB as part of routine investigation or staging for prostate cancer
* Aged 18-80 years
* BMI between 19.5 and 35 kg/m2
* Smokers and non-smokers

Exclusion Criteria:

* Those regularly taking 5α-reductase inhibitors or testosterone replacement medicines
* Those on warfarin treatment
* Those diagnosed with diabetes
* Those diagnosed with or suspected to be high-risk for human immunodeficiency virus (HIV) and/or hepatitis
* Those allergic to any of the ingredients of the broccoli soups
* Those taking dietary supplements or herbal remedies which may affect the study outcome. Please note that some supplements may not affect the study and this will be assessed on an individual basis
* Those that are unable to understand English or give informed consent
* Parallel participation in another research project that involves dietary intervention
* Any person related to or living with any member of the study team

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Sulphate level | Biopsy on a single occasion at ≥ 4 weeks
  Sulphate levels will be measured in biopsy tissue samples from both prostate and adipose (fat) tissues.

SECONDARY OUTCOMES:
ADP | Biopsy on a single occasion at ≥ 4 weeks
  Adenosine diphosphate (ADP) levels will be measured in biopsy tissue samples from both prostate and adipose (fat) tissues.
Redox status of phosphatase proteins | Biopsy on a single occasion at ≥ 4 weeks
  The redox status of phosphatase proteins, including the tumour suppressor PTEN will be assessed in biopsy tissue samples from the prostate gland.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Coode-Bate J, Sivapalan T, Melchini A, Saha S, Needs PW, Dainty JR, Maicha JB, Beasy G, Traka MH, Mills RD, Ball RY, Mithen RF. Accumulation of Dietary S-Methyl Cysteine Sulfoxide in Human Prostate Tissue. Mol Nutr Food Res. 2019 Oct;63(20):e1900461. doi: 10.1002/mnfr.201900461. Epub 2019 Sep 11. PMID 31410992